CLINICAL TRIAL: NCT05607693
Title: A Multi-Center, Open- Label, Single-Arm Phase 1 QT/QTc Study of SHR3680 in Subjects With Castration-Resistant Prostate Cancer
Brief Title: A SHR3680 QT/QTc Study on Castration-Resistant Prostate Cancer Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR3680-I-QTc
Record Dates: First submitted 2022-10-12; First posted 2022-11-07 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Castration-Resistant Prostate Cancer

STUDY DESIGN:
Intervention Model Description: Multiple dose of SHR3680 will be administered
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR3680 (Experimental)
  Interventions: Drug: SHR3680 tablets

INTERVENTIONS:
Drug: SHR3680 tablets — Subjects start taking SHR3680 tablets 240 mg/dose/day orally on an empty stomach on D1, and the timing of administration daily should be consistent when possible.

SUMMARY:
The purpose of this study is to determine whether daily treatment with SHR3680 affects the ventricular repolarization in participants with Castration-Resistant Prostate Cancer (CRPC).

ELIGIBILITY:
Inclusion Criteria:

1. Male between 18 years to 75 years of age;
2. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
3. Expected survival of at least 6 months;
4. Histologically or cytologically confirmed adenocarcinoma of the prostate without indication of neuroendocrine or small cell features; nonmetastatic castration-resistant prostate cancer (NM-CRPC) or metastatic castration-resistant prostate cancer (mCRPC) ;
5. Be surgically or medically castrated and if treated with a gonadotropin releasing hormone analog (ie, patient who has not undergone bilateral orchiectomy), then this therapy must have been initiated at least 4 weeks prior to Day 1 and must be continued throughout the study;
6. Castrated level of testosterone at screening (≦ 50 ng/dL or 1.73 nmol/L);
7. Organ function level must meet the following requirements (blood transfusion or hematopoietic growth factor therapy was not received within 2 weeks before blood test):

   * ANC≧1.5×109/L；
   * PLT≧80×109/L；
   * Hb≧90 g/L；
   * TBIL≦1.5×ULN；
   * ALT and AST≦2.5×ULN；
   * BUN and Cr≦1.5×ULN；
   * GFR≧60ml/min/1.73m2；
8. 12-lead ECG: heart rate ≥ 50 beats/min, PR interval within 110-220 ms (including both ends), QTc interval corrected according to Fridericia 's criteria (QTcF) < 470 msec. Left ventricular ejection fraction (LVEF) ≥ 50% by echocardiography;
9. Able to complete the study as required by the protocol;
10. Sign the informed consent before the trial, and fully understand the trial content, process and possible adverse reactions.

Exclusion Criteria:

1. Washout period of any previous anti-tumor therapy (including radiotherapy, chemotherapy, surgery, molecular targeted therapy, immunotherapy, androgen receptor antagonists, CYP-17 inhibitors, 5α-reductase inhibitors, estrogen, progesterone drugs, etc.) to the of the first dose of this study drug is < 4 weeks;
2. Plan to receive any other anti-tumor therapy during the treatment phase in this trial;
3. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 4 weeks;
4. Known brain metastases;
5. history of epilepsy, or past medical history of disease that can induce seizures (including transient ischemic attack history, cerebral stroke (except cerebral ischemic lesions only found in imaging test), brain trauma with disturbance of consciousness requiring hospitalization) within 12 months before the first dose of the study drug;
6. past medical history of the following diseases within 6 months before screening: myocardial infarction, severe/unstable angina, NYHA class II-IV cardiac insufficiency, ≥ Grade 2 sustained arrhythmia (graded based on NCI CTCAE 5.0), heart failure, grade II-III atrioventricular block, complete left bundle branch block, atrial fibrillation of any grade, coronary/peripheral artery bypass graft or stenting, cerebrovascular accident (including transient ischemic attack), pulmonary embolism, deep vein thrombosis;
7. Inability to swallow, chronic diarrhea and intestinal obstruction, or the presence of multiple other factors affecting drug administration and absorption;
8. Patients with active HBV or HCV infection (HBV copy number ≥ 104 copies/mL, HCV copy number ≥ 103 copies/mL);
9. Patients with immunodeficiency disease history (including HIV test positive, other acquired or congenital immunodeficiency diseases) or organ transplantation history;
10. Patients who are unwilling to take protocol-specified contraceptive measures throughout the study treatment period and within 3 months after the last dose;
11. History of significant hypersensitivity, intolerance, or allergy to any drug compound or known allergy to SHR3680 or the excipients;
12. Excessive smoking (≥ 5 cigarettes/day) within 6 months before screening or smoking within 48 h before the first dose, or positive at nicotine screening test, and can't abstain from smoking during the study; History of drug abuse, positive at drug abuse screening, or history of any drug use in the past 6 months;
13. History of alcoholism or regular alcohol consumption within 6 months before screening, that is, drinking more than 14 units of alcohol per week (1 unit = 360 mL of beer with 5% alcohol or 45 mL of spirits with 40% alcohol or 150 mL of wine with 12% alcohol) or drinking within 48 h before the first dose, or positive at alcohol breath test on the day of admission, or unable to abstain during the study;
14. Subjects who took any vitamins, health products or herbal medicine within 14 days before dosing;
15. Subjects who took any beverage or food containing grapefruit, xanthine, caffeine, or alcohol within 48 hours before dosing; strenuous exercise; or other factors which affect drug absorption, distribution, metabolism, excretion, etc;
16. Abnormal coagulation function (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or APTT > 1.5 ULN), bleeding tendency or on thrombolytic therapy;
17. Patients with implantable pacemaker and automatic implantable cardioverter defibrillator;
18. Personal or family history of long QT syndrome;
19. Use of Medications that prolong QT/QTc interval or with risk of torsades de pointes (TdP) within 7 days prior administration of study drug;
20. Significant history or clinical manifestation of concomitant diseases or other situations that put serious hazards to the patient' s safety, or affect the patient 's completion of the study, as determined by the Investigator.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2024-11-05 (Estimated); Study Completion 2024-11-05 (Estimated)

PRIMARY OUTCOMES:
Delta QTc Fridericia (QTcF) | Day -1 and Day 1 and Day 17
  Mean change from baseline in QTcF as measured based on triplicate electrocardiograms extracted from continuous 12-lead Holter monitor recordings after study drug intake.
Concentration-delta QTcF relationship | Day -1 and Day 1 and Day 17
  Relationship between SHR3680 plasma concentration and delta QTcF based on linear-mixed effect model.

SECONDARY OUTCOMES:
Electrocardiographic parameters Delta PR | Day -1 and Day 1 and Day 17
  A change from time-matched baseline measurements in PR interval will be determined on Day -1, Day 1 and Day 17.
Electrocardiographic parameters Delta RR | Day -1 and Day 1 and Day 17
  A change from time-matched baseline measurements in RR interval will be determined on Day -1, Day 1 and Day 17.
Electrocardiographic parameters Delta QRS | Day -1 and Day 1 and Day 17
  A change from time-matched baseline measurements in QRS interval will be determined on Day -1, Day 1 and Day 17.
Electrocardiographic parameters Delta QTc Bazett (QTcB) | Day -1 and Day 1 and Day 17
  Mean change from baseline in QTcB as measured based on triplicate electrocardiograms extracted from continuous 12-lead Holter monitor recordings after study drug intake.
Electrocardiographic parameters T-wave morphology | Day -1 and Day 1 and Day 17
  Number and percentage of participants with changes from baseline
Electrocardiographic parameters U-wave morphology | Day -1 and Day 1 and Day 17
  Number and percentage of participants with changes from baseline
Incidence and severity of AE/SAE/AESI (rated based on CTCAE v5.0) | Day-1, Day 1 to Day 18
  Participants will be monitored for safety during the Screening and Treatment Phases, and up to 30 days after the last dose of study drug. From the end of treatment phase onward collection of AE will be limited to Grade 3 or higher, all SAE and AESI from the remainder of the study.
Pharmacokinetic parameter area under the plasma drug concentration-time curve (AUC) from time 0 to 24 hours | Day 1-2 and Day 17-18
Pharmacokinetic parameter maximum concentration observed (Cmax) | Day 1-2 and Day 17-18
Pharmacokinetic parameter time to reach Cmax (tmax) | Day 1-2 and Day 17-18
Pharmacokinetic parameter minimum observed plasma concentration at steady-state (Cmin,ss) | Cmin,ss will only be collected on Day 17
Pharmacokinetic parameter accumulation ratio（Rac） | Day 1-2 and Day 17-18

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital of Tianjin, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided